CLINICAL TRIAL: NCT03362060
Title: A Phase 1b Study of Safety and Immune Response to PVX-410 Vaccine Alone and in Combination With Pembrolizumab in HLA-A2+ Patients With Metastatic Triple Negative Breast Cancer (TNBC)
Brief Title: PVX-410 Vaccine Plus Pembrolizumab in HLA-A2+ Metastatic Triple Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Steven J Isakoff, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-328
Record Dates: First submitted 2017-11-27; First posted 2017-12-05 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Triple Negative Breast Cancer; Metastatic Breast Cancer
Keywords: Triple Negative Breast Cancer; Vaccine; Immunotherapy; PD-1 Inhibitor; Metastatic Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — pembrolizumab; PVX-410 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PVX-410 (Experimental): * PVX-410 vaccine at W0, 1, 2, 3, 4, and 5 followed by booster PVX-410 vaccine doses at W10 and 28
  * Pembrolizumab will be administered every 3 weeks intravenously starting with week 1
  Interventions: Drug: Pembrolizumab; Biological: PVX-410

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a monoclonal antibody checkpoint inhibitor that blocks a protein in T-cells cells called PD-1, which then allows these cells and other parts of the immune system to attack tumors
  Other Names: Keytruda
Biological: PVX-410 — PVX-410 is a type of vaccine composed of 4 9-amino acid peptides that may help the immune system stimulate immunity against cancer cells

SUMMARY:
This research study is studying immunotherapy as a possible treatment for metastatic Triple Negative Breast Cancer (TNBC) in participants who are HLA-A2+.

The drugs involved in this study are:

* PVX-410
* Pembrolizumab
* Hiltonol
* Montanide

DETAILED DESCRIPTION:
This research study is a Phase Ib clinical trial, which tests the safety of an investigational drug combination and also tries to better understand how the investigational intervention affects the body.

"Investigational" means that the FDA (the U.S. Food and Drug Administration) has not approved the combination of PVX-410 and pembrolizumab as a treatment regimen for this specific disease.

The FDA has not approved PVX-410 as a treatment for any disease. PVX-410 is a type of vaccine that may help the immune system stimulate immunity against the cancer cells.

The FDA has not approved pembrolizumab for this specific disease but it has been approved in the United Sates for other types of cancer.

Pembrolizumab is a drug that may treat cancer by working with the immune system. The immune system is the body's natural defense against disease. The immune system sends types of cells throughout the body to detect and fight infections and diseases, including cancer. For some types of cancer, the immune cells do not work as they should and are prevented from attacking the tumors. Pembrolizumab is thought to work by blocking a protein in the cells called Programmed Death-1 (PD-1), which then allows these cells and other parts of the immune system to attack tumors.

In this research study, the investigators are studying the body's immune response to the PVX-410 study vaccine in combination with pembrolizumab. This study will help researchers understand if the vaccine and pembrolizumab can work together to help the body's immune system recognize and treat triple negative breast cancer. The investigators are also studying the safety of the PVX-410 together with the pembrolizumab

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for the study.
* Female aged ≥18 years on the day of signing informed consent.
* HLA A2+ by deoxyribonucleic acid (DNA) sequence analysis (by history with documentation or as part of this study).
* Histopathological diagnosis of metastatic or inoperable locally advanced TNBC that meets the following criteria:

  --Triple negative defined as Estrogen Receptor (ER)<1%, Progesterone Receptor (PR)<1%, and Human Epidermal Growth Factor Receptor 2 (HER2) negative according to American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines by local testing according to institutional standards.
* For tumors with equivocal interpretation of receptor status (e.g., ER/PR ≥1% "weak" or "faint" staining), the Principal Investigator will have final determination of triple-negative status. For tumors with discrepant receptor results between 2 or more biopsies (including metastatic and/or early stage biopsies), the Principal Investigator will have final determination of triple negative status, but in general the most recent biopsy can be used for eligibility purposes. If receptor testing is not available on a metastatic biopsy, the primary tumor test result is acceptable.
* Metastatic or inoperable locally advanced disease is defined as either: histologically confirmed metastatic breast cancer by biopsy; or locally advanced breast cancer that, in the opinion of the treating physician, is not amenable to curative intent surgical resection; or, radiological or clinical evidence suggestive and supportive of metastatic disease without a documented metastatic biopsy, provided the patient has a prior diagnosis of TNBC that otherwise meets the eligibility criteria.

  --Ductal, lobular, mixed, or metaplastic histology.
* Measurable disease, as determined by RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (see Appendix section 16.1)
* At least one line of prior systemic therapy for metastatic or recurrent breast cancer (there is no limit to the number of prior therapies).
* Adequate normal organ and marrow function within 10 days of planned treatment initiation, as defined below:

Hematologic

* Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L without transfusion or erythropoietin dependency (within 7 days of assessment)
* Absolute neutrophil count (ANC) ≥1.5x10^9/L (≥1500 per mm3)
* Platelet count ≥100x109/L (≥100,000 per mm3) Renal
* Serum creatinine ≤1.5 x the upper limit of normal (ULN) OR measured or calculated creatinine clearance ≥60 mL/min for patients with creatinine levels >1.5 x institutional Upper Limit of Normal (ULN) (calculated per institutional standard). (Glomerular filtration rate can be used in place of creatinine or creatinine clearance.) Hepatic
* Serum bilirubin ≤1.5 x institutional ULN OR direct bilirubin ≤ ULN for patients with total bilirubin levels >1.5 x ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤2.5 x institutional ULN OR ≤5 x ULN for patients with known liver metastases.
* Albumin ≥2.5 mg/dL Coagulation
* International normalized ratio (INR) or prothrombin time (PT) ≤1.5 x ULN, unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
* Activated partial thromboplastin time (aPTT) ≤1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Other
* Lactate Dehydrogenase (LDH) ≤1.5 x institutional ULN

  * Willing to provide archived tissue for correlative studies. If no archived sample is available the patient will still be eligible.
  * Negative virology/serology for human immunodeficiency virus (HIV)-1, HIV-2, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) DNA.
  * Either of non-reproductive potential (i.e., post-menopausal by history of age ≥50 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, history of bilateral tubal ligation, or history of bilateral oophorectomy) OR must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
  * If of childbearing potential (i.e., does not meet criteria for non-reproductive potential above), willing to use 2 methods of birth control, or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study treatment
  * Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations, including follow-up

Exclusion Criteria:

* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study treatment.
* Previous enrollment in the present study.
* Mucinous or tubal histology or other good prognosis histology.
* Known hypersensitivity to any component of PVX-410, Hiltonol®, Montanide, pembrolizumab, or excipients.
* Receipt of the last dose or treatment of anti-cancer chemotherapy, radiotherapy, surgery, endocrine therapy, targeted therapy, biologic therapy, or tumor embolization ≤2 weeks (4 weeks for any monoclonal Antibody (mAb), 6 weeks for nitrosoureas or mitomycin C) prior to first dose of study treatment, or has not recovered (i.e., to ≤Grade 1 or Baseline) from clinically significant Adverse Events (AEs) due to these previously administered agents.

  * Patients with ≤Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Subjects with other irreversible toxicity (e.g., hearing loss) or reversible toxicity (e.g. alopecia) that is not reasonably expected to be exacerbated by the investigational product and is not expected to interfere with study participation may be included.
  * If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Received a live vaccine within 30 days of planned start of study therapy.

  --Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Ongoing or planned systemic anti-cancer therapy or radiation therapy.
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the pre-screening or screening visit through 120 days after the last dose of study treatment.
* Has a known history of active Tuberculosis (Bacillus Tuberculosis).
* History of allogeneic organ transplant.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for management of brain metastases for at least 7 days prior to study treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Known history of non-infectious pneumonitis that required steroids or any evidence of active pneumonitis.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* History or current evidence of any other condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-12-12 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Immune Response following treatment with PVX-410 in combination with pembrolizumab | 3 years
  The fold activation of T cells from blood of treated patients at week 10 compared to baseline

SECONDARY OUTCOMES:
Late Immune response after treatment with PVX-410 and pembrolizumab | 3 years
  The fold activation of T cells from blood of treated patients at week 28 compared to baseline.
Incidence of treatment emergent adverse events (safety and tolerability) of PVX-410 in combination with pembrolizumab | 3 years
  Number of patients who develop treatment emergent adverse events according to the Common Toxicity Criteria of Adverse Events (CTCAE) version 4.0
Progression Free Survival | 3 years
  The median time from study enrollment to disease progression of all treated participants.
Overall Survival | 3 years
  The median time from study enrollment of all participants until death of all treated participants.
Response rate | 3 years
  The rate of RECIST defined responses (complete and partial response).

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Isakoff, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No